CLINICAL TRIAL: NCT03065283
Title: Effects of Diaphragm-releasing Techniques on the Lumbar Spine and Diaphragmatic Function in Healthy Women: a Randomized Clinical Trial
Brief Title: Effects of Diaphragm-releasing Techniques on the Lumbar Spine and Diaphragmatic Function in Healthy Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Ceara (Other)
Responsible Party: Principal Investigator, Pedro Olavo de Paula Lima, University professor of physiotherapy course Federal University of Ceará, Universidade Federal do Ceara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: POdePLima2
Record Dates: First submitted 2017-02-06; First posted 2017-02-27 (Actual); Results first posted 2020-04-07 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Healthy Individuals

STUDY DESIGN:
Intervention Model Description: The sample was randomly divided by electronic draw in two groups, the intervention group (GI), where two techniques were performed, one for diaphragmatic release and another for relaxation of the diaphragm pillars. In the control group (CG) the same techniques were applied, but in a placebo form.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diaphragmatic release (Active Comparator): The stretching of the peripheral fibers of the diaphragm
  Interventions: Procedure: Diaphragm lift; Procedure: Relaxation of the diaphragm pillars
- Diaphragmatic release control (Placebo Comparator): In both placebo techniques, only the light touching of the contacts of the volunteers' skin
  Interventions: Procedure: Diaphragm lift; Procedure: Relaxation of the diaphragm pillars

INTERVENTIONS:
Procedure: Diaphragm lift — The purpose is to generate the stretch of the peripheral fibers of the diaphragm, being performed with the patient in the supine position and the physiotherapist standing on the patient's head and Pulling the Your costal arch In the cephalic direction, for one minute, twice
  Other Names: Diaphragmatic release 1
Procedure: Relaxation of the diaphragm pillars — Second technique aims to promote the rhythmic stretching of the double psoas diaphragm pillars, being performed with The patient in the ventral position and the therapist standing at his side placing the ulnar border of his cephalic hand on the last ribs and his caudal hand flattened in front of the popliteal fossa of the popliteal fossa, stretching was done for one minute
  Other Names: Diaphragmatic release 2

SUMMARY:
The aim of this study was to evaluate the immediate effects of diaphragmatic release techniques on posterior chain flexibility and lumbar spine amplitude. Respiratory muscle strength and chest cavity mobility in healthy women.

DETAILED DESCRIPTION:
The aim of this study was to evaluate the immediate effects of diaphragmatic release techniques on posterior chain flexibility and lumbar spine amplitude; Respiratory muscle strength and chest cavity mobility in healthy women. This is an intervention study with a randomized controlled trial design. The randomized study in two groups, the Intervention Group in which two diaphragmatic release techniques were performed and the Control Group where two placebo techniques were applied in 75 participants between 18 and 35 years of age. For intragroup analysis the paired Student t test was used, comparing the outcomes before and after the intervention and for intergroup analysis the independent Student t test.

ELIGIBILITY:
Inclusion Criteria:

* sedentary female participants
* aged between 18 and 35 years.

Exclusion Criteria:

* those with cardiovascular, respiratory obstructive or restrictive disease
* smokers and ex-smokers
* who were or were submitted to speech therapy less than a year ago
* those with postural deviation type scoliosis

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marizeiro DF, Florencio ACL, Nunes ACL, Campos NG, Lima POP. Immediate effects of diaphragmatic myofascial release on the physical and functional outcomes in sedentary women: A randomized placebo-controlled trial. J Bodyw Mov Ther. 2018 Oct;22(4):924-929. doi: 10.1016/j.jbmt.2017.10.008. Epub 2017 Oct 25. PMID 30368336

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: none declare
Period: Overall Study
Arm/Group | Diaphragmatic Release | Diaphragmatic Release Control
Started | 50 | 25
Completed (Outcomes were measured at baseline and after intervention. There was no dropoput of sample.) | 50 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diaphragmatic Release | Diaphragmatic Release Control | Total
Number analyzed (Participants) | 50 | 25 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.24 (2.86) | 21.12 (2.12) | 21.18 (2.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 25 | 75
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Thoracic Mobility
Description: Thoracic mobility was measued with a tape as an evaluation tool.
Time Frame: baseline and immediately post-intervention
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Diaphragmatic Release | Diaphragmatic Release Control
Number analyzed (Participants) | 50 | 25
cm
  baseline | 2.87 (0.93) | 2.78 (1.08)
  post-intervention | 3.47 (1.00) | 2.86 (0.99)
Statistical Analysis 1: Comparison: Diaphragmatic Release vs Diaphragmatic Release Control; A paired t-test was used for intragroup analysis, and an independent Student's t-test was used for intergroup analysis. Data are represented in mean between-group difference with a 95% CI, and analysis was by intention to treat; Test type: Equivalence — p< or = 0.05; p = 0.05, t-test, 2 sided; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [-0.38 to 0.57]

2. Other Pre Specified Outcome: Amplitude of Motion of the Lumbar Spine
Description: Tape measure was used as an evaluation tool.
Time Frame: baseline and immediately post-intervention
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Posterior Chain Flexibility
Description: Tape measure was used as an evaluation tool.
Time Frame: baseline and immediately post-intervention
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Maximum Respiratory Pressure
Description: manovacuometer was used as an evaluation tool.
Time Frame: baseline and immediately post-intervention
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Diaphragmatic Release | Diaphragmatic Release Control
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/25
Other Adverse Events (participants affected / at risk) | 0/50 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No